CLINICAL TRIAL: NCT05698706
Title: High Intensity Focused Ultrasound (HIFU) Treatment of Basal Cell Carcinoma: Efficacy and Safety
Brief Title: High Intensity Focused Ultrasound (HIFU) Treatment of Basal Cell Carcinoma
Acronym: HIFU-BCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jacek Calik (Other)
Responsible Party: Sponsor-Investigator, Jacek Calik, Managing Director, Old Town Clinic, Poland
Organization: Old Town Clinic, Poland (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFU-BCC-2023-1
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Basal Cell Carcinoma
Keywords: Skin cancer; HIFU; BCC; Dermatology; High Intensity Focused Ultrasound; Dermoscopy
MeSH Terms: conditions — Carcinoma, Basal Cell; Skin Neoplasms

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- De-novo BCC with thickness not more than 2.0 mm (Experimental): Areas with de-novo BCC of thickness not more than 2.0 mm (as confirmed by ultrasound imaging or histopathological examination) will be treated by high intensity focused ultrasound
  Interventions: Device: TOOsonix System ONE-M

INTERVENTIONS:
Device: TOOsonix System ONE-M — Selected BCC sites will be treated using high intensity focused ultrasound

SUMMARY:
The overall objective of the study is to evaluate the safety and efficacy of treatment of Basal Cell Carcinoma (BCC) using a new modality based on high-intensity focused ultrasound (HIFU). BCC is the most common type of skin cancer in Europe, Australia and the US. It accounts for more than 75% of all skin cancer cases in those regions. There are currently more the 14000 BCC cases registrations in Poland every year, and occurrences on a global scale are counted in several millions per year. Given the trend of aging population those numbers will only increase with time. Finding new and more effective treatment methods are therefore highly relevant from both a clinical and socioeconomic perspective. The investigational device used in the study is a system capable of making controlled and targeted thermo-mechanical treatment of small intradermal volumes containing e.g. BCC cells, but without inflicting damage to the surrounding tissue.

The investigation involves an evaluation of the safety and efficacy profile 3 months after a single few-minute treatment. Subsequent follow-up of secondary endpoints is done every third month until the end of the study one year after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of each gender aged 18 years or older at the time of informed consent. There is no upper limit of age.
* Subjects who have received oral and written study information, accepted participation and signed the informed consent document.
* Subjects who are willing and mentally and physically capable to understand and follow the treatment and follow-up schedule including post-treatment care instructions.
* Subjects who are willing to have photographs and images taken of the treated lesions to be used anonymously or coded in evaluations and publications.
* Subjects, who have histologically and clinically verified basal cell carcinoma cancer of thickness not more 2.0 mm measured by ultrasound imaging or histopathological examination.

Exclusion Criteria:

* Subjects who are less than 18 years at the time of informed consent.
* Subject is pregnant or lactating at time of first treatment
* Subjects with extensive, invasive or advanced skin cancer when another method in use such as radiotherapy or Mohs' surgery has priority and offers the patient better opportunity of cure.
* Cancers on anatomical sites where the ultrasound probe cannot be adapted for anatomical reasons
* Any systemic disease that according to investigator's assessment may interfere with the spontaneous course of a skin cancer.
* Any condition predisposing to treatment-related adverse effects or complications from the ultrasound treatment.
* Subjects with abnormal scar formation
* Subjects with impaired wound healing
* Subjects with any other acute or chronic condition which, in the opinion of the investigator, could interfere with the conduct of the study
* Subjects undergoing immunosuppressive treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2022-12-14 (Actual); Primary Completion 2025-05-14 (Estimated); Study Completion 2025-05-14 (Estimated)

PRIMARY OUTCOMES:
Cure rate | 3 months
  Frequency of complete clearance of BCC after HIFU treatment. Binary output: yes/no
Severity of short term adverse events | 3 months
  Safety profile after treatment of basal cell carcinoma measured on a 4-point severity score ranging from No side effects (score 0) to Severe side effects (score 3)

SECONDARY OUTCOMES:
Severity of adverse events | 12 months
  Any objective adverse effect or event, local or systemic, related to the treatment and the investigational device (wound and course of wound healing, scar formation, instrumental hazards) measured at 6, 9 and 12 months. Measured on a 4-point severity score ranging from No side effects (score 0) to Severe side effects (score 3)
Cure rate | 12 months
  Frequency of complete clearance of BCC after HIFU treatment measured at 6, 9, 12 months after HIFU treatment. Binary output: yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Calik, MD, PhD, Principal Investigator — Old Town Clinic
Locations (1):
- Old Town Clinic, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bove T, Zawada T, Serup J, Jessen A, Poli M. High-frequency (20-MHz) high-intensity focused ultrasound (HIFU) system for dermal intervention: Preclinical evaluation in skin equivalents. Skin Res Technol. 2019 Mar;25(2):217-228. doi: 10.1111/srt.12661. Epub 2019 Jan 8. PMID 30620418
- [Background] Soegaard S, Aarup V, Serup J, Bove T, Zawada T, Jessen A, Poli M. High-frequency (20 MHz) high-intensity focused ultrasound system for dermal intervention: A 12-week local tolerance study in minipigs. Skin Res Technol. 2020 Mar;26(2):241-254. doi: 10.1111/srt.12786. Epub 2019 Sep 20. PMID 31541524
- [Background] Serup J, Bove T, Zawada T, Jessen A, Poli M. High-frequency (20 MHz) high-intensity focused ultrasound: New Treatment of actinic keratosis, basal cell carcinoma, and Kaposi sarcoma. An open-label exploratory study. Skin Res Technol. 2020 Nov;26(6):824-831. doi: 10.1111/srt.12883. Epub 2020 Jun 17. PMID 32557832
- [Background] Calik J, Zawada T, Bove T. Treatment of superficial benign vascular tumors by high intensity focused ultrasound: Observations in two illustrative cases. J Cosmet Dermatol. 2022 Aug;21(8):3371-3379. doi: 10.1111/jocd.14682. Epub 2021 Dec 17. PMID 34921489
- [Background] Calik J, Migdal M, Zawada T, Bove T. Treatment of Seborrheic Keratosis by High Frequency Focused Ultrasound - An Early Experience with 11 Consecutive Cases. Clin Cosmet Investig Dermatol. 2022 Jan 28;15:145-156. doi: 10.2147/CCID.S348106. eCollection 2022. PMID 35125879
- See also: Website of Old Town Clinic — https://oldtownclinic.pl/en/